CLINICAL TRIAL: NCT03079336
Title: Design Development in Randomized Clinical Trials - Psychological Treatment in Generalized Anxiety
Brief Title: Implementation of Psychological Treatment in Generalized Anxiety
Acronym: IMPLEMENT2_0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PP00P1_163702
Record Dates: First submitted 2017-01-12; First posted 2017-03-14 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: Randomized controlled design development; Translational Research; Psychological Interventions; Contextual Model of Psychotherapy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- State of the art (SOTA) check-in phase (Experimental): The therapists will apply the usual SOTA check-in phase lasting between 5 and 10 minutes, as recommended in the preexisting guideline including reviewing progress in self-help and agenda setting (Zinbarg et al., 2006).
  Interventions: Behavioral: Implementation - SOTA; Behavioral: Mastery your Anxiety and Worry (MAW)
- Prolonged focus on subtle changes (Experimental): Based on the robust findings that over 90% of the patients will experience subtle changes, the therapists will extend the above mentioned check-in phase by systematized focus for 7 to 20 minutes capitalizing on small and subtle changes and exceptions.
  Interventions: Behavioral: Implementation - Prolonged focus on changes; Behavioral: Mastery your Anxiety and Worry (MAW)

INTERVENTIONS:
Behavioral: Implementation - SOTA — The implementation of an evidence-based treatment is largely principle-based - allowing considerable therapeutic flexibility in determining and timing of different treatment aspects. In this condition progress, subtle changes and sudden gains may be an explicit topic and there is no restraint to avoid such topics. However, the therapists are not obligated to take a systematized focus on potential subtle changes and they may use the timing of the sessions to involve the patients into the other tasks of therapy.
  Arms: State of the art (SOTA) check-in phase
Behavioral: Implementation - Prolonged focus on changes — Systematized sequence of exploration of subtle changes at a prolonged check-in phase: (1) the precise change situation, (2) related emotional states, (3) related helpful thoughts and self-verbalizations, (4) reinforcement of generalized self-efficacy and treatment motivation, (5) benefit for the upcoming session goals (Flückiger, Grosse Holtforth, et al. 2013, 2014).
  Arms: Prolonged focus on subtle changes
Behavioral: Mastery your Anxiety and Worry (MAW) — In the present study, the MAW-packet will be applied within a usual 16-session individual therapy format and up to 3 further booster sessions.
  The session format of 50-60 minute usually consists of (a) a check-in phase of 5 to 15 minutes that includes a patients welcoming, reviewing self-help and agenda setting, (b) a working phase around 35-45 minutes that focuses on the previously agreed session goals, (c) a feedback phase of 5 to 10 minutes that summarizes the session and previews the upcoming self-help assignment.
  Other Names: Cognitive Behavioral Therapy

SUMMARY:
Pragmatic randomized controlled trial (expected N = 80) of cognitive-behavioral therapy (CBT) to contrast two psychotherapeutic implementation strategies (State-of-the-Art welcome phase vs. prolonged focus on sudden changes). Blinded allocation of implementation strategy for patients; open label for therapists (no blinding possible), randomized allocation for patients, therapist allocation via ABAB-design (crossed-therapist design). Post treatment self-reported outcome will be measured based on a latent outcome factor (i. e. "outcome composite").

DETAILED DESCRIPTION:
State of research. The proposed trial has a common theme, i.e., the understanding of the enduring efficacy of psychological treatments in individuals who suffer from general anxiety disorder (GAD). There is meta-analytic evidence that bona fide psychotherapy is an effective treatment for GAD, but also for individuals that suffers from anxiety and depression. Nonetheless, in spite of the empirical evidence of the overall efficacy, there is a lack of randomized controlled studies that systematically investigate the therapists' variability (i. e. therapist effects) within the very same treatment protocol. The development of study designs to investigate potential health professional effects along treatment effects is a general claim for human interventions. This protocol includes one of the very first process-outcome trials in GAD that systematically examine theory-based patients' and therapists' characteristics simultaneously using longitudinal multilevel methodology.

Along with investigating therapist and patient characteristics, two methods for timing the check-in phase at the beginning of each session will be compared by keeping constant the standardized treatment manual for patients with GAD: (a) prolonged focus on subtle changes check-in condition lasting from 7 to 20 minutes and (b) a state of the art (SOA) check-in phase lasting from 5 to 10 minutes. To address the nested data structure, therapists will be allocated by a single-subject ABAB-design. A total of 80 patients (40 participants in each of the two conditions) with a primary GAD diagnosis will be treated by 20 advanced cognitive-behavioral therapy trainees at the psychotherapy outpatient clinic in the department of psychology at the university of Zürich.

Relevance. (a) Study population. GAD is a neglected disorder in the Swiss mental health system. GAD is associated with personal suffering, a reduced quality of life, and high economic costs. (b) Design development. Systematic integration of potential therapist effects is a neglected aspect in many areas of evidence-based human interventions (inside but also outside of psychological interventions). (c) Treatment development. Evidence-based treatments are usually far from being fully efficacious. There is a debate about innovative research agendas and how to foster the efficacy of such treatments. (d) Experimental process-outcome research. There is a need for future research to investigate theory-based therapist effects and in-session timing within rigorous experimental process-outcome research designs to better understand the factors involved in therapeutic change (e.g. http://www.nature.com/news/therapy-deficit-1.11477).

ELIGIBILITY:
Inclusion Criteria:

1. fulfill the diagnostic criteria for GAD based on the structured interview for DSM,
2. are 18 years of age or older,
3. Mastery of German language
4. are seeking out a cognitive-behavioral therapy (CBT) for GAD at the outpatient clinic (Attenhoferstrasse 9) of the Institute for Psychology of the University of Zürich
5. Informed consent as documented by signature

Exclusion Criteria:

1. Acute Suicidal Ideation (BDI Suicide item > 1 or suicidal ideation in the telephone interview)
2. Currently taking a psychotic or bipolar disorder medication, or
3. Currently receiving treatment from a professional psychotherapist/psychiatrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months treatment completion of a latent 5-facet, self-report outcome-factor | Baseline, treatment completion after 6 months (16 sessions)
  Latent factor of the below-mentioned 5 self-report questionnaires (outcome composite)

OTHER OUTCOMES:
Penn State Worry Questionnaire [PSWQ] | Baseline, treatment completion after 6 months (16 sessions)
  Self-report worry inventory (Meyer et al., 1990)
Beck Anxiety Inventory [BAI] | Baseline, treatment completion after 6 months (16 sessions)
  Self-report anxiety inventory (Beck et al., 1988)
Beck Depression Inventory II [BDI-II] | Baseline, treatment completion after 6 months (16 sessions)
  Self-report depression inventory (Beck et al., 1996)
Short version of the Symptom Check List [SCL-9] | Baseline, treatment completion after 6 months (16 sessions)
  Self-report symptom severity index (Klaghofer & Brähler, 2001)
Short version of the Resource Self-Report Questionnaire [RES] | Baseline, treatment completion after 6 months (16 sessions)
  Self-report resource inventory (Troesken & Grawe, 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Flueckiger, Prof Dr., Principal Investigator — Department of Psychology, University of Zürich
Locations (1):
- Department of Psychology, University of Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fluckiger C, Visla A, Wolfer C, Hilpert P, Zinbarg RE, Lutz W, Grosse Holtforth M, Allemand M. Exploring change in cognitive-behavioral therapy for generalized anxiety disorder-A two-arms ABAB crossed-therapist randomized clinical implementation trial. J Consult Clin Psychol. 2021 May;89(5):454-468. doi: 10.1037/ccp0000639. Epub 2021 Apr 8. PMID 33829819
- [Derived] Visla A, Allemand M, Fluckiger C. Within- and between-patients associations between self-efficacy, outcome expectation, and symptom change in cognitive behavioral therapy for generalized anxiety disorder. J Clin Psychol. 2023 Jan;79(1):86-104. doi: 10.1002/jclp.23407. Epub 2022 Jul 4. PMID 35781807
- [Derived] Visla A, Constantino MJ, Fluckiger C. Predictors of change in patient treatment outcome expectation during cognitive-behavioral psychotherapy for generalized anxiety disorder. Psychotherapy (Chic). 2021 Jun;58(2):219-229. doi: 10.1037/pst0000371. PMID 34410791
- [Derived] Fluckiger C, Horvath AO, Brandt H. The evolution of patients' concept of the alliance and its relation to outcome: A dynamic latent-class structural equation modeling approach. J Couns Psychol. 2022 Jan;69(1):51-62. doi: 10.1037/cou0000555. Epub 2021 Jul 1. PMID 34197151
- [Derived] Fluckiger C, Wolfer C, Held J, Hilpert P, Rubel J, Allemand M, Zinbarg RE, Visla A. How to customize a bona fide psychotherapy for generalized anxiety disorder? A two-arms, patient blinded, ABAB crossed-therapist randomized clinical implementation trial design [IMPLEMENT 2.0]. BMC Psychiatry. 2018 Apr 3;18(1):86. doi: 10.1186/s12888-018-1666-2. PMID 29614982